CLINICAL TRIAL: NCT00675662
Title: TrimTots Pre-school Obesity Prevention Programme
Brief Title: Trim Tots Pre-school Obesity Prevention Programme
Acronym: TrimTots
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Child Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 07NT14
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2015-09

CONDITIONS: Overweight; Obesity
Keywords: Obesity; overweight; BMI; ifestyle; diet; nutrition; physical activity; pre-school; toddlers; children; Prevention of overweight and obesity in pre-school children
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Stratification by angiotensin converting enzyme (ACE) genotype
  Interventions: Behavioral: Lifestyle intervention
- 2 (Placebo Comparator): Waiting list controls
  Interventions: Behavioral: waiting list control

INTERVENTIONS:
Behavioral: Lifestyle intervention — Lifestyle intervention with Trim Tots pre-school programme.
  Arms: 1
Behavioral: waiting list control — waiting list control
  Arms: 2

SUMMARY:
Randomised controlled trial of a lifestyle intervention programme for mothers and children aged 1-5 years aimed at prevention of overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Children who are currently overweight/obese or at increased risk of becoming so and their mother or usual carer.

Ages: 12 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2008-04; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Body Mass index | 12 months

SECONDARY OUTCOMES:
Cardiovascular (CV) disease risk factors | 12 months
Physical activity (accelerometry) | 12 months
Motor co-ordination (ABC battery). | 12 months
Motor co-ordination (ABC battery). Behaviour (general and dietary). | 12 months
CV fitness (heart rate variability). | 12 months
Waist circumference | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lanigan, Principal Investigator — Institute of Child Health
Locations (1):
- Institute of Child Health, 30 Guilford Street, London, United Kingdom

REFERENCES:
- [Background] Summerbell CD, Waters E, Edmunds LD, Kelly S, Brown T, Campbell KJ. Interventions for preventing obesity in children. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD001871. doi: 10.1002/14651858.CD001871.pub2. PMID 16034868
- [Background] Flynn MA, McNeil DA, Maloff B, Mutasingwa D, Wu M, Ford C, Tough SC. Reducing obesity and related chronic disease risk in children and youth: a synthesis of evidence with 'best practice' recommendations. Obes Rev. 2006 Feb;7 Suppl 1:7-66. doi: 10.1111/j.1467-789X.2006.00242.x. PMID 16371076
- See also: Obesity guidance on the prevention, identification, assessment and management of overweight and obesity in adults and children. National Institute for Health and Clinical Excellence. — http://guidance.nice.org.uk/CG43/niceguidance/word/English